CLINICAL TRIAL: NCT00309972
Title: A Randomized Phase III Trial of Sequential Chemotherapy Followed By Radical Radiotherapy Versus Concurrent Chemo-Radiotherapy Followed by Chemotherapy in Patients With Inoperable Stage III Non-Small Cell Lung Cancer and Good Performance Status
Brief Title: Cisplatin, Vinorelbine, and Radiation Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer That Cannot Be Removed By Surgery
Acronym: SOCCAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000465629; C11922/A4558 (Other Grant/Funding Number: Cancer Research UK); 13746987 (Other: ISRCTN); EU-20602 (Other: UCL CTC); 2004-001920-19 (EudraCT Number)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential arm (SEQ) (Active Comparator): Four cycles of cisplatinum/vinorelbine given in a 21 day cycle followed by radical radiotherapy, 55 Gy in 20 once daily fractions in four weeks (2.75 Gy/day).
  Interventions: Drug: Control arm (SEQ):
- Experimental arm (CON) (Experimental): Concurrent chemo-radiotherapy [55 Gy in 20 daily fractions in 4 weeks (2.75 Gy/day) with cisplatinum given concurrently with fractions 1-4 and 16-19, and vinorelbine prior to fractions 1, 6, 15 and 20] followed by two cycles of cisplatinum/vinorelbine.
  Interventions: Drug: Experimental arm (CON):

INTERVENTIONS:
Drug: Control arm (SEQ): — Four cycles of cisplatinum/vinorelbine given in a 21 day cycle followed by radical radiotherapy, 55 Gy in 20 once daily fractions in four weeks (2.75 Gy/day).
  Arms: Sequential arm (SEQ)
Drug: Experimental arm (CON): — concurrent chemo-radiotherapy [55 Gy in 20 daily fractions in 4 weeks (2.75 Gy/day) with cisplatinum given concurrently with fractions 1-4 and 16-19, and vinorelbine prior to fractions 1, 6, 15 and 20] followed by two cycles of cisplatinum/vinorelbine.
  Arms: Experimental arm (CON)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether giving combination chemotherapy followed by radiation therapy is more effective than giving combination chemotherapy together with radiation therapy followed by more chemotherapy in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying combination chemotherapy followed by radiation therapy to see how well it works compared to combination chemotherapy combined with radiation therapy followed by more chemotherapy in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with stage III non-small cell cancer treated with chemotherapy comprising cisplatin and vinorelbine ditartrate (CV) followed by radical radiotherapy versus concurrent CV chemoradiotherapy followed by CV chemotherapy.

Secondary

* Compare the progression-free survival of patients treated with these regimens.
* Compare the local progression-free survival (local control).
* Compare the hematological, pulmonary, esophageal, and neurological toxicities.
* Compare the response.
* Compare the quality of life.
* Compare the cost-effectiveness.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to clinically important factors. Patients are randomized to 1 of 2 treatment arms.

* Arm I (sequential treatment): Patients receive cisplatin IV over 2 hours on day 1 and vinorelbine ditartrate IV over 5-10 minutes on days 1 and 8. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Beginning in week 15, patients undergo radiotherapy 5 days a week for 4 weeks.
* Arm II (concurrent treatment): Patients undergo radiotherapy as in arm I beginning in week 1. Patients receive cisplatin IV over 2 hours on days 1-4 and vinorelbine ditartrate IV over 5-10 minutes on days 1 and 8. Chemotherapy repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, monthly for 6 months, and then at each follow-up visit.

After completion of study treatment, patients are followed periodically.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 508 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage III non-small cell lung cancer (NSCLC)

  * Patients with stage IIIB disease must not have a pleural effusion that is cytologically proven to be malignant
* Inoperable disease
* Disease must be able to be encompassed within a radical radiotherapy treatment volume

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* Life expectancy > 3 months
* Patient considered able to tolerate platinum-based chemotherapy and radical radiotherapy
* Glomerular filtration rate ≥ 60 mL/min
* WBC > 3,000/mm³
* Absolute neutrophil count > 1,500/mm³
* Hemoglobin > 10.0 g/dL

  * Patients with hemoglobin between 10 and 12 g/dL at randomization require a blood transfusion to ensure hemoglobin > 12 g/dL before starting radiotherapy
* Platelet count > 100,000/mm³
* FEV_1 ≥ 1.0 L or DLCO (transfer factor) ≥ 50% of predicted
* Alkaline phosphatase ≤ 1.5 times upper limit of normal (ULN)
* Gamma-glutamyl-transferase < 1.5 times ULN
* Transaminases ≤ 1.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* No medically unstable conditions (e.g., unstable diabetes, uncontrolled arterial hypertension, infection, hypercalcemia, or ischemic heart disease)
* Not pregnant or nursing
* Fertile patients must agree to use effective contraception
* Negative pregnancy test
* No other previous or current malignant disease likely to interfere with protocol treatment or comparisons

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-12; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Treatment related mortality (any cause) | from randomization till death

SECONDARY OUTCOMES:
Hematological, pulmonary, esophageal, and neurological toxicities | From randomisation to the first 6 months
Quality of life | at baseline, every 3 weeks for the first 6 months, then 3 monthly until 2 years, 6 monthly until 3 years, and annually thereafter
Cost effectiveness | at baseline, every 3 weeks for the first 6 months, then 3 monthly until 2 years, 6 monthly until 3 years, and annually thereafter
Overall survival and progression-free survival. | Overall Survival is the time between date of randomisation and date of death of any cause. Progression-free survival will be calculated from the date of randomisation to the date of first clinical evidence of progressive disease, or death.
Local progression-free survival (local control) | From the date of randomisation to the date of first clinical evidence of progressive disease at the primary site, or death
Response | proportion of patients in each treatment group whose best response in the first 6 months from randomisation is complete or partial will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Maguire, MD, Study Chair — Clatterbridge Centre for Oncology
Locations (1):
- Clatterbridge Centre for Oncology, Merseyside, England, United Kingdom